CLINICAL TRIAL: NCT02044029
Title: A SINGLE CENTER, LONGITUDINAL, NON-DRUG STUDY TO ASSESS THE ABILITY OF MUSCLE IMAGING AND OF MOTOR FUNCTION MEASURE (MFM) TO DETECT CHANGES IN DISEASE PROGRESSION IN AMBULANT SPINAL MUSCULAR ATROPHY (SMA) PATIENTS AS COMPARED TO AGE-MATCHED HEALTHY CONTROLS
Brief Title: Ability of Muscle Imaging and Motor Function Measure (MFM) to Detect Changes in Disease Progression in Ambulant Spinal Muscular Atrophy Patients Compared to Healthy Volunteers.
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: BE29037
Record Dates: First submitted 2014-01-16; First posted 2014-01-23 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer, Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples taken at screening and at week 24 from patients with spinal muscular atrophy (SMA).

GROUPS / COHORTS (2):
- Age- and gender-matched controls
- Patients with spinal muscular atrophy

SUMMARY:
This non-drug, single center, 24-week, longitudinal study in ambulant spinal muscular atrophy (SMA) patients and in age- and gender-matched healthy volunteers will assess the detection of disease progression by magnetic resonance imaging (MRI) and the Muscle Function Measure (MFM) test.

Each participant will be evaluated in three testing sessions: at baseline, at Week 12 and at Week 24. Both patients and volunteers will undergo MRI scans. Patients will additionally undergo testing of motor function and have blood samples taken for Survival of the Motor Neuron (SMN) genes, proteins and mRNA analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, aged >/= 10 years at screening
* For SMA patients: Confirmed clinical diagnosis of 5q-autosomal recessive SMA, ambulant at time of screening, and prefereably without spinal cord fixation

Exclusion Criteria:

* Previous (3 months or less) or concomitant participation in any other therapeutic trial
* Known or suspected cancer
* Other chronic disease or inadequate renal, liver, or heart function
* Contraindications for MRI scans, including but not limited to: claustrophobia, pacemaker, artifical heart valves, cochlear implants, presence of foreign metal objects in the body, intracranial vascular clips, etc. Any contraindications to MRI found on a standard radiography scan.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Ambulant patients with spinal muscular atrophy (SMA) and age- and gender-matched healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Differences in quantitative muscle MRI based on fat content and T2 values | At baseline, Week 12 and Week 24
Disease progression, assessed through the Motor Function Measure test | At baseline, Week 12 and Week 24

SECONDARY OUTCOMES:
Disease progression, assessed with the 6-minute Walk Test. | At baseline, Week 12 and Week 24
Levels of Survival of Motor Neuron (SMN) RNA | At baseline and Week 24
Levels of SMN proteins | At baseline and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Basel, Switzerland